CLINICAL TRIAL: NCT04473586
Title: Validation Protocol Spartan Cube CYP2C19- Method Comparison
Brief Title: Spartan Cube CYP2C19 Method Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spartan Bioscience Inc. (Industry)
Collaborators: Mount Sinai Services (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: VNV-00229
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Genotyping Techniques
Keywords: Method Comparison; CYP2C19

STUDY DESIGN:
Intervention Model Description: All subjects will experienced the same number of buccal and saliva samples collected. This means all subjects will participate in Arm 1 and have materials collected at the same time in the event they are enrolled in arm 2.
  Based on enrollment numbers and their immediate genotype, it will be determined at that time if the subject will participate in the second arm of the study.
Who Masked: Participant, Investigator
Masking Description: Bi-directional sequencing results and Spartan results will not be shared with participants. The investigator will not see the bi-directional sequencing results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sample tested in less than one-hour (Other): Buccal samples will be collected and analyzed on the Spartan Cube CYP2C19 System immediately (<1hr). The Spartan Cube CYP2C19 results will be compared with bi-directional sequencing results generated by a third part from a saliva sample collected from the same subject.
  Interventions: Device: Spartan Cube CYP2C19 System
- Samples tested greater than 24 hours (Other): Buccal samples will be collected, stored and then analyzed on the Spartan Cube CYP2C19 System greater than 24 hours after collection. The Spartan Cube CYP2C19 results will be compared with bi-directional sequencing results generated by a third part from a saliva sample collected from the same subject.
  Interventions: Device: Spartan Cube CYP2C19 System

INTERVENTIONS:
Device: Spartan Cube CYP2C19 System — Using buccal material, determine the genotype of the *2, *3 and *17 SNPs of the CYP2C19 gene on the Spartan Cube CYP2C19 System.

SUMMARY:
The aim of the study is to demonstrate concordance (percent agreement) between results produced by the Spartan CYP2C19 system and bi-directional sequencing. In addition, this study will evaluate the concordance of buccal samples stored prior to running on the Spartan Cube CYP2C19 system and bi-directional sequencing.

DETAILED DESCRIPTION:
Sample holding time - two parts

1. Sample tested in less than one-hour

   a.In the first part, buccal samples will be collected from subjects and tested using the Spartan Cube CYP2C19 system. These samples will be run immediately (within 1 h) after collection from the subject (<1 h sample holding time). All results will be compared to bi-directional sequencing to determine percent agreement.
2. Sample tested greater than 21 hours a.In the second part (sample holding portion), samples will be tested using the Spartan Cube CYP2C19 product. These samples will be run after storage at ambient temperature. All results will be compared to bi-directional sequencing to determine the percent agreement.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will provide buccal samples and a saliva sample who have not eaten drank or smoked in the past 30 minutes.

Exclusion Criteria:

* Participants who have eaten drank or smoked in the past 30 minutes prior to collection.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
% Agreement of test results generated on the Spartan Cube CYP2C19 System and bidirectional sequencing | Through study completion; anticipated to be less than 4 months
  Determine % agreement across all tests conducted and bi-directional sequencing results

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Ahmed, PhD, Principal Investigator — Spartan Bioscience Inc.
Locations (1):
- Mount Sinai Services, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No